CLINICAL TRIAL: NCT03969160
Title: Neural Activations During Imaginal Exposure in Individuals Fearful of Spiders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017/419
Record Dates: First submitted 2019-05-24; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Individuals With Fear of Spiders
Keywords: Imaginal exposure; brain imaging; mental imagery
MeSH Terms: interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaginal exposure (Experimental): The experimental procedure consists of imaginal exposure to mental imagery of phobic and neutral stimuli, prompted through recorded verbal instructions. Participants' repeat the experimental procedure one week later in a follow-up session. Brain imaging data is only collected during day 1
  Interventions: Behavioral: Imaginal exposure

INTERVENTIONS:
Behavioral: Imaginal exposure — Imaginal exposure to mental imagery of phobic and neutral stimuli

SUMMARY:
This study explores the brain basis of imaginal exposure, a widely used psychological treatment technique. Specifically, this study uses functional magnetic resonance imaging to examine brain areas activated during imaginal exposure, in individuals fearful of spiders. Physiological responses and subjective fear experienced during imaginal exposure are also assessed.

The primary aim of this study is to explore differences in neural activity during exposure to phobic, compared to neutral, mental imagery. The study will focus primarily on exploratory whole brain analyses, but will also include regions of interest analyses on brain areas previously associated with imaginal exposure. The experimental procedure consists of repeated exposure to mental imagery, i.e. imagery of short durations, including either highly emotion-provoking or neutral content, prompted by verbal instructions. A secondary aim is to explore the effects of repeated exposure to mental imagery, used during the experimental procedure, on subjective fear and physiological responses.

DETAILED DESCRIPTION:
Results will elucidate if neural activity to phobic imagery differs from activity associated with the production of mental imagery per se. Findings will also increase our general understanding of the neural basis of imaginal exposure treatments.

ELIGIBILITY:
Inclusion Criteria:

* Significant fear of spiders

Exclusion Criteria:

* Current psychiatric disorder other than spider phobia
* Substance abuse
* Neurological disease
* Psychological treatment or psychotropic medication within six months
* Magnetic resonance imaging contradiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level dependent contrast (BOLD-signal) | Day 1
  BOLD-signal is assessed using functional magnetic resonance imaging.
Physiological response during exposure to mental imagery | Day 1
  Skin-conductance responses are used as a measure of physiological response.

SECONDARY OUTCOMES:
Physiological response during exposure to mental imagery | Follow-up (one week after day 1)
  Skin-conductance responses are used as a measure of physiological response.
Differences in physiological response during exposure to mental imagery, during day 1 compared to the follow-up session. | Difference between day 1 and the follow-up session (one week after day 1)
  Skin-conductance responses are used as a measure of physiological response.
Ratings of subjective fear participants' expect to experience during exposure to mental imagery | Day 1
  Scale: 0-100; no fear at all - extreme fear.
Ratings of subjective fear experienced during exposure to mental imagery | Day 1
  Scale: 0-100; no fear at all - extreme fear. Fear ratings are completed immediately after the imaginal exposure experimental procedure
Spielberger State-Trait Anxiety Inventory (STAI-S) | Day 1
  STAI-S is a self-rated questionnaire included to assess state-anxiety experienced during exposure. High scores indicate high levels of state anxiety (range, total score: 20 - 80).
Differences in ratings of subjective fear during exposure to mental imagery, during day 1 compared to the follow-up session. | Difference between day 1 and the follow-up session (one week after day 1)
  Scale: 0-100; no fear at all - extreme fear.
Vividness of mental imagery | Day 1
  Vividness of mental imagery of phobic stimuli (scale: 1-5; no image at all - image as clear and vivid as real life).
Vividness of mental imagery | Follow-up (one week after day 1)
  Vividness of imagery of phobic stimuli (scale: 1-5; no image at all - image as clear and vivid as real life).
Differences in vividness of mental imagery, during day 1 compared to the follow-up session. | Difference between day 1 and the follow-up session (one week after day 1)
  Vividness of imagery of phobic stimuli (scale: 1-5; no image at all - image as clear and vivid as real life).
Difficulties in emotion regulation scale (DERS) | Day 1
  DERS is a self-rated questionnaire, included to explore potential relations between imaginal exposure and difficulties in emotion regulation. High scores indicate more difficulties in emotion regulation (range, total score: 36 - 180)

OTHER OUTCOMES:
Spider Phobia Questionnaire (SPQ) | Recruitment
  SPQ is a self-rated questionnaire assessing fear of spiders. A high score in SPQ (>19) is required for inclusion in the study.
Spielberger State-Trait Anxiety Inventory (STAI-T) | Day 1
  STAI-T is a self-rated questionnaire assessing trait anxiety and is included to describe the sample in terms of anxiety proneness. High scores indicate higher levels of trait anxiety (range, total score: 20 - 80)
Number of intrusive mental imagery of phobic stimuli | 7 days, starting on day 1.
  Number of intrusive mental images of phobic stimuli recorded by participants in a diary, daily (morning, afternoon, evening and night) for 7 days. This measure is included as a manipulation check.
Demand questions | Day 1
  Two questions asking participants' to appreciate the emotional impact of producing mental imagery versus focusing on the verbal aspects of phobic situations used in the experimental procedure. This measure is included as a manipulation check.
The Plymouth Sensory Imagery Questionnaire (Psi-Q) | Day 1
  The Psi-Q is a self-rated measure of vividness of imagery across different sensory modalities. Higher scores indicate higher levels of vividness (range, total score 0 - 70).

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Uppsala University Hospital - Akademiska sjukhuset, Uppsala
  - Uppsala University, Departement of Psychology, Uppsala